CLINICAL TRIAL: NCT06871917
Title: The Relation of Maternal Iron Deficiency and/or Iron Deficiency Anemia to Neonatal Hemoglobin Concentration and Iron Stores
Brief Title: Maternal Iron Deficiency and/or Iron Deficiency Anemia to Neonatal Hemoglobin Concentration and Iron Stores
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Naglaa A. Ali, assistant lecturer at family medicine department AUH, Assiut University
Other Study IDs: FAMAssiutU
Record Dates: First submitted 2025-03-07; First posted 2025-03-12 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Relation, Mother-Child
Keywords: anemia iron deficiency iron stores

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
study the relationship between maternal iron deficiency (ID) and/or iron deficiency anemia (IDA) to neonatal hemoglobin concentration and iron stores at birth

DETAILED DESCRIPTION:
Iron deficiency is a common micronutrient deficiency in pregnant women specially in developing countries as increasing demands on maternal iron stores as consequences of expansion of maternal red blood cell mass and the requirement of the developing fetus.

The relationship between maternal iron stores and fetal iron extraction has received considerable attention as iron deficiency places neonates at high risks for cognitive, motor, social-emotional, and neurodevelopmental problem. moreover, requirement of iron is high for rapid growth and differentiation of the fetus and thus a well-balanced iron hemostasis is required. This balance can be threatened in neonates born to iron compromised mothers.

Some studies have suggested that the fetus reflects maternal iron stores, but this concept is still being debated as few other studies show contrasting results, majority of studies have been done in developed countries. To draw the consensus regarding the result, more studies needed to clarify the effect of maternal iron status on fetal stores are required. Proper understanding of the relationship between maternal and neonatal iron indices will help in formulating protocols that is required to improve the maternal and neonatal outcomes, so investigating the effect maternal iron on fetal iron indices can be of great value, so that early intervention to prevent or reverse the adverse effect of iron deficiency on development issues much before iron deficiency becomes sever can be instituted.

ELIGIBILITY:
Inclusion Criteria:

* All pregnant women and their infant pairs who have given consent to participate.
* Mothers Age: 21-40 years' old.
* Term infants (37-42 weeks of gestation) with birth weight ≥2500 g born to mothers who had an uncomplicated normal singleton vaginal delivery or caesarian section delivery was included.

Exclusion Criteria:

* Mothers with a history of antepartum hemorrhage, pre-mature labor pain, high-risk pregnancy (eg. history of trauma and severe infection during pregnancy), severe hyperemesis, pre-eclampsia severe anemia requiring blood transfusion, and any chronic medical illnesses as: gestational diabetes, hypertension, hypothyroidism, epilepsy, liver disease, renal disease cardiorespiratory disease, immunodeficiency syndrome, and hematological (other causes of anemia)
* infants who suspected with congenital and/or chromosomal anomalies and pathological jaundice, also multiple pregnancy was excluded from the study.
* Mothers withdrew from given a written consent will be excluded from the study.

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study will include all pregnant women meet the inclusion criteria and their infant pairs at the time of delivery.
Sampling Method: Probability Sample
Enrollment: 370 (Estimated)
Dates: Start 2025-06-08 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation the effect of maternal iron deficiency (ID) and/or iron deficiency anemia (IDA) to fetal haemoglobin concentration and fetal iron stores. | 2 years
  evaluation the correlation between ID and IDA in maternal and neonatal samples

SECONDARY OUTCOMES:
-Prevalence of maternal iron deficiency and/or iron deficiency anemia at birth in our community. | 2 years
  finding the prevalence of ID and/or IDA in pregnant mother
-Effect of maternal iron deficiency and/or iron deficiency anemia on early neonatal outcome . | 2 years
  exploring early neonatal outcomes after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Dalia G. Mahran, prof, Study Director — prof of public health and community medicine, Faculty of medicine, Assuit university
Locations (1):
- Naglaa Ali Ali, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Krafft A, Huch R, Breymann C. Impact of parturition on iron status in nonanaemic iron deficiency. Eur J Clin Invest. 2003 Oct;33(10):919-23. doi: 10.1046/j.1365-2362.2003.01244.x. PMID 14511365
- [Background] Bentley DP. Iron metabolism and anaemia in pregnancy. Clin Haematol. 1985 Oct;14(3):613-28. PMID 3907911
- [Background] Mei Z, Cogswell ME, Looker AC, Pfeiffer CM, Cusick SE, Lacher DA, Grummer-Strawn LM. Assessment of iron status in US pregnant women from the National Health and Nutrition Examination Survey (NHANES), 1999-2006. Am J Clin Nutr. 2011 Jun;93(6):1312-20. doi: 10.3945/ajcn.110.007195. Epub 2011 Mar 23. PMID 21430118
- [Background] Scholl TO. Iron status during pregnancy: setting the stage for mother and infant. Am J Clin Nutr. 2005 May;81(5):1218S-1222S. doi: 10.1093/ajcn/81.5.1218. PMID 15883455
- [Background] Lozoff B. Iron deficiency and child development. Food Nutr Bull. 2007 Dec;28(4 Suppl):S560-71. doi: 10.1177/15648265070284S409. PMID 18297894
- [Background] Delaney KM, Guillet R, Fleming RE, Ru Y, Pressman EK, Vermeylen F, Nemeth E, O'Brien KO. Umbilical Cord Serum Ferritin Concentration is Inversely Associated with Umbilical Cord Hemoglobin in Neonates Born to Adolescents Carrying Singletons and Women Carrying Multiples. J Nutr. 2019 Mar 1;149(3):406-415. doi: 10.1093/jn/nxy286. PMID 30770543
- [Background] Bernhardt GV, Jhancy M, Shivappa P, Bernhardt K, Pinto JRT. Relationship between maternal and cord blood iron status in women and their new born pairs. Vol. 14, Biomedical and Pharmacology Journal. 2021. p. 317-22.